CLINICAL TRIAL: NCT00618462
Title: Cognitive Behavioral Treatments for Pathological Gambling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01MH060417-09 (NIH); R01MH060417-09 (NIH); 04-428 (Other: Institutional Review Board); DATR A2-AIR
Record Dates: First submitted 2008-02-15; First posted 2008-02-20 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Gambling
Keywords: Cognitive Behavioral Therapy; Pathological Gambling
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy; Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive psychoeducation therapy plus case management and a referral to Gamblers Anonymous.
  Interventions: Behavioral: Psychoeducation therapy; Behavioral: Case management; Behavioral: Gamblers Anonymous (GA)
- 2 (Experimental): Participants will receive cognitive behavioral therapy plus contingency management and a referral to Gamblers Anonymous.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT); Behavioral: Contingency management (CM); Behavioral: Gamblers Anonymous (GA)
- 3 (Experimental): Participants will receive cognitive behavioral therapy and a referral to Gamblers Anonymous.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT); Behavioral: Gamblers Anonymous (GA)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — CBT will include weekly 50-minute sessions for 8 weeks. The sessions will focus on learning skills to cope with urges to gamble and developing alternatives to gambling.
  Arms: 2; 3
Behavioral: Contingency management (CM) — CM will provide incentive, such as a gift certificate to a store or restaurant, for completing activities not related to gambling. Participants and their therapists will decide upon two potential alternative activities to gambling during each therapy session.
  Arms: 2
Behavioral: Psychoeducation therapy — Psychoeducation therapy will include weekly 50-minute therapy sessions for 8 weeks. The sessions will focus on education about gambling and related problems.
  Arms: 1
Behavioral: Case management — Case management will assist participants in obtaining additional services from the community as needed.
  Arms: 1
Behavioral: Gamblers Anonymous (GA) — All participants will be referred to GA, a support group of people who are recovering from gambling addiction, and will be encouraged to attend meetings.

SUMMARY:
This study will determine the effectiveness of three different treatment strategies in reducing gambling behaviors in pathological gamblers.

DETAILED DESCRIPTION:
Pathological gambling is a chronic disorder in which a person is unable to control the urge to gamble. People who are pathological gamblers constantly think about gambling, and they may feel restless when not able to gamble. A pathological gambler's addiction to the thrill of gambling may lead to serious relationship, career, and debt problems. The number of pathological gamblers in the United States is steadily growing, leading to significant financial, psychological, and public health consequences. However, studies examining the effectiveness of treatments for pathological gamblers are limited. Forms of psychotherapy, such as cognitive behavioral therapy (CBT), and addiction support groups comprise some of the commonly used treatments for pathological gamblers. This study will compare the effectiveness of three different treatment strategies, including psychoeducation therapy plus case management, CBT, and CBT plus contingency management (CM), in reducing gambling behaviors and other problems related to pathological gambling.

Participation in this study will last 2 years. All potential participants will undergo an initial screening that will include questions about gambling behaviors and related problems and psychiatric, medical, social, legal, and substance abuse history. Eligible participants will be referred to Gambler's Anonymous (GA) and will be randomly assigned to one of three treatment groups. All participants will attend a 50-minute session of their assigned treatment each week for 8 weeks. They will also be encouraged to attend GA meetings during treatment.

* Group 1 participants will receive psychoeducation therapy plus case management. Therapy sessions will include education about gambling and related problems. The case management component of treatment will offer help with obtaining additional services from the community as needed.
* Group 2 participants will attend CBT sessions, which will include learning about the triggers that lead to gambling, developing alternatives to gambling, and avoiding relapse after stopping gambling.
* Group 3 participants will receive CM in addition to CBT, as described above. The CM component of treatment will encourage participants to partake in activities unrelated to gambling by awarding vouchers, such as a gift certificate to a store or restaurant, to participants for completing the alternative activities.

Gambling, substance use, and psychosocial problems will be assessed at pretreatment and Months 2, 6, 9, 12, 18, and 24 follow-up evaluations. Participants will also be asked to identify at least one person who is aware of their gambling problem and whom they regularly contact. Researchers will interview the contact person by phone at pretreatment and Months 2, 6, 12, and 24. The interview will include questions about the participant's gambling behaviors, personal relationships, legal status, use of health care and mental health services, and any possible change of contact information.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00158314

http://clinicaltrials.gov/show/NCT00118391

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for pathological gambling
* At least two gambling episodes in the 60 days prior to study entry

Exclusion Criteria:

* Inability to read English at the 5th grade level (as assessed by the Slosson Oral Reading Test)
* Uncontrolled psychiatric conditions (e.g., active suicidal intention, psychosis, bipolar disorder, or current alcohol or drug dependence other than nicotine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2004-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Addiction Severity Index (ASI) gambling severity scores | Measured at pretreatment and Months 2, 6, 9, 12, 18 and 24 follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M. Petry, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States